CLINICAL TRIAL: NCT00531115
Title: Multicentre, Single-arm, Phase II Study to Evaluate Safety and Efficacy of Cetuximab in Combination With Oxaliplatin and Capecitabine (XELOX) for 12 Weeks Followed by Maintenance Treatment With Cetuximab Plus Capecitabine as First-line Treatment in Elderly Patients With Metastatic Colorectal Cancer.
Brief Title: Phase II Study to Evaluate Safety and Efficacy of Cetuximab in Combination With XELOX for 12 Weeks Followed by Maintenance Treatment With Cetuximab Plus Capecitabine as First-line Treatment in Elderly Patients With Metastatic Colorectal Cancer.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: According to the study design, in the first step the number of responses was lower than the number required (< 7).
Sponsor: Spanish Cooperative Group for the Treatment of Digestive Tumours (TTD) (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TTD-06-05; EudraCT Nº: 2006-007062-11
Record Dates: First submitted 2007-09-17; First posted 2007-09-18 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Metastatic Colorectal Cancer
Keywords: metastatic colorectal cancer; elderly patients; cetuximab, oxaliplatin, capecitabine
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: cetuximab 5mg/ml

INTERVENTIONS:
Drug: cetuximab 5mg/ml — Weekly administration of Cetuximab (initial infusion of 400 mg/m2 for 120 minutes followed by subsequent maintenance doses of 250 mg/m2 for 60 minutes) Oxaliplatin. 130 mg/m2 every three weeks. on day 1 for 4 cycles Capecitabine. 1000 mg/m2 twice daily (2.000 mg/m2 total daily dose) or 750 mg/m2 if Cl Cr=30-50 ml/min (1500 mg/m2 total daily dose) for two weeks (on days 1 to 14) followed by one week of rest (on days 15 to 21).
  The patients will receive 4 cycles of cetuximab plus combination chemotherapy administered every 3 weeks in order to achieve a noticeable response. Then, oxaliplatin treatment will be stopped after a maximum of 4 infusions to prevent appearance of neuropathy and then followed by capecitabine 2 weeks out of 3, and cetuximab weekly as maintenance treatment.

SUMMARY:
The purpose of this study is to determine confirmed objective response rate to combination therapy with cetuximab plus XELOX for 4 cycles followed by maintenance treatment with cetuximab plus capecitabine as first line treatment in elderly patients with metastatic colorectal cancer

DETAILED DESCRIPTION:
* This open-label, non-controlled, multicentre, phase II study will recruit 53 elderly patients with diagnosis of metastatic colorectal cancer.
* All patients will receive 4 cycles of treatment with cetuximab plus XELOX followed by cetuximab plus capecitabine as maintenance therapy until progression of disease, occurrence of unacceptable toxicity to the study drugs, or withdrawal of consent by the patient.
* The planned duration of a cycle is 3 weeks.
* Cetuximab therapy will not be delayed for chemotherapy-related toxicity and vice versa. If patients benefit from combination therapy, but develop unacceptable intolerance to oxaliplatin and/or capecitabine, cetuximab may be continued in combination with the other chemotherapy drug and/or as a single agent. In case of cetuximab intolerance, patients should continue with chemotherapy treatment until progression disease.
* Evaluations:

  * Efficacy data (response rate, progression-free survival, duration of response and survival) and safety data will be collected. The investigators will assess responses to treatment.
  * When the treatment is stopped either because of disease progression or occurrence of unacceptable toxicity, the patients will enter a follow-up period where the progression-free survival, the subsequent lines of treatment and the survival data will be collected every 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent before any study related activities are carried out
* Men and women >= 70 years.
* Histologically confirmed diagnosis of CRC.
* Non-resectable and/or non-operable metastatic colorectal carcinoma.
* Presence of at least one lesion by two-dimensional measurement; index lesions should not be in a region with previous irradiation.
* Availability of tumor tissue for immunohistochemical analysis
* Karnofsky functional status >= 80% at the time of enrollment in the study.
* Life expectancy greater than 3 months.
* Patients will not have received chemotherapy for advanced or metastatic disease. Patients with the following characteristics will be included: 1. Recurrence after neoadjuvant and/or adjuvant treatment with 5-fluorouracil/folinic acid or capecitabine +/- radiotherapy with disease-free interval > 12 months following conclusion of treatment. 2. Recurrence after surgical and/or radiotherapy treatment without adjuvant systemic treatment. 3. De novo diagnosis of disease.
* Proper hematological, renal and hepatic function,

Exclusion Criteria:

* Documented or suspected cerebral and/or leptomeningeal metastases.
* Surgery (excluding biopsy for diagnosis) and/or radiotherapy during the 4 weeks prior to inclusion in the study.
* Chronic, concomitant systemic immunotherapy, chemotherapy, or hormonal treatment for cancer.
* Prior administration of monoclonal antibodies, EGFR signal transduction inhibitors or EGFR-targeted treatment.
* Participation in another clinical trial with medication in the past 30 days
* Prior participation in a study in which treatment with cetuximab may be assigned (whether or not treatment with cetuximab is received).
* Prior malignant tumor in the past 5 years, except for history of adequately treated basal cell skin cancer or pre-invasive cervical cancer .
* Lack of physical integrity of the upper gastrointestinal tract or malabsorption syndrome or history of inflammatory intestinal disease, acute or subacute intestinal occlusion or other disease which could alter drug absorption.
* Evidence of grade 3 or 4 allergic reaction to any treatment components or other fluoropyrimidines.
* Clinically relevant peripheral neuropathy.
* Clinically significant coronary artery disease or history of myocardial infarction in the last 12 months or high risk of decompensation of heart failure or arrhythmia.
* Serious active infections (requiring intravenous antibiotics), including active tuberculosis and diagnosed HIV.
* Known abuse of alcohol/drugs.
* Legal incapacity or limited legal capacity.
* Any medical or psychological disorder which, in the opinion of the investigator, does not allow the patient to conclude the study or sign the informed consent.
* Patients catalogued as delicate or "frail" for compliance with any of the following criteria

  * Dependence in one or more activities of daily life according to the Katz Activity of Daily Living (ADL) scale.
  * 3 or more comorbid entities based on evaluation of the presence of the following processes: congestive heart failure; valvular heart disease; coronary artery disease; obstructive or restrictive chronic pulmonary disease; cerebrovascular disease; peripheral neuropathies; chronic renal failure; hypertension; diabetes; concomitant neoplasms; collagen vascular diseases; and incapacitating arthritis.
  * Presence of geriatric syndromes: moderate-severe dementia; delirium in situation of stress (urinary or respiratory infection, angina or drugs); moderate-severe depression that interferes with usual activity of patient; frequent falls (3 or more per month); lack of care (Who could help him or her in the event of an emergency?); urinary incontinence in the absence of stress, infection, diuretics or prostatic hyperplasia; fecal incontinence in the absence of diarrhea or laxatives; osteoporotic fractures of long bones or vertebral crush.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 28 (Actual)
Dates: Start 2007-11; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Confirmed objective response rate | 2007-2009

SECONDARY OUTCOMES:
Disease control, Time to progression, progression-free survival,Time to treatment failure,Determine time to onset of response, Duration of response, Overall survival, To determine biologic prognostic factors | 2007-2009
Treatment safety | 2007-2009

CONTACTS AND LOCATIONS:
Overall Officials: Javier Sastre, Study Chair — H. Clinico San Carlos. Madrid. Spain
Locations (1):
- Spanish Cooperative Group for Gastrointestinal Tumour Therapy, Madrid, Spain

REFERENCES:
- See also: Related Info — http://www.ttdgroup.org